CLINICAL TRIAL: NCT01154049
Title: Phase 1 Study to Evaluate the Safety of the Vaccine Prepared sm14 Against Schistosomiasis
Brief Title: Study to Evaluate the Safety of the Vaccine Prepared sm14 Against Schistosomiasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Financiadora de Estudos e Projetos (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: sm14-CT001P1
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Schistosomiasis
Keywords: Schistosomiasis; Vaccine; sm14
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): 3 doses of the vaccine, on days 0, 30 and 60.
  Interventions: Biological: sm14 antigen plus adjuvant GLA

INTERVENTIONS:
Biological: sm14 antigen plus adjuvant GLA — Healthy adults will receive 3 doses of the vaccine, on days 0, 30 and 60.

SUMMARY:
This is a phase I, open-label, single arm trial, which aims to assess the safety of the vaccine prepared sm14 in healthy subjects. The product immunogenicity will be evaluated by conducting serology (anti-sm14 antibodies) and testing of cellular response to the antigen by the method ELI-SPOT. Each participant will remain in the study for approximately 4 months. The total study duration is 10 months, considering a period of 6 months for inclusion. Will be included in the study subjects male and female, between 18 and 49 years, that manifest their will to participate in the research by signing an Informed Consent Form. Eligible population for the study are subjects who do not present at screening significant changes in renal, cardiac and liver functions, complete blood count, clotting, present no acute or chronic illnesses, are not in the chronic use of any medication, do not have HIV infection or other immunodeficiency. Pregnant or breastfeeding women will not be included. Volunteers will receive three doses of vaccine prepared sm14, in doses containing 50 mcg of the antigen, associated with adjuvant GLA-SE at a dose of 10 mcg, with an interval of 30 days between each application. Twenty volunteers will be included in the study. This is a convenience sample, established for the first test of the product in humans, for the initial safety assessment.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 49 years.
* Available for follow-up throughout the study period (approximately 120 days).
* Ability to understand and sign the informed consent form (IC).
* HIV serology negative
* Absence of helminth infections in general (nematodes, cestodes and trematodes, among which Schistosoma mansoni) at the inclusion in the study.
* Patients who has not chronic use or have not used in the past 45 days any medication, except trifling as nasal saline and vitamins.
* Be in good health without significant medical history.
* Screening physical examination without clinical significant abnormalities.
* Screening laboratory tests without significant abnormalities according to normal standards and the evaluation of investigators.
* Additional criteria for females of childbearing potential: Negative pregnancy test at screening; consistent use of contraceptive methods (male or female condom, diaphragm, IUD and oral contraceptives or "patches").

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Use of cytotoxic or immunosuppressive drugs in the last six months, except for spray nasal corticosteroids for allergic rhinitis or topical corticosteroids for uncomplicated dermatitis.
* Immunoglobulin use 60 days prior to vaccination.
* Use of any type of vaccine 30 days prior to vaccination.
* Plan to receive any other vaccine during the period of participation in the study (four months)
* Use any type of investigational medication in a period of 30 days prior to vaccination
* Use of allergy shots with antigens within 14 days prior to vaccination.
* Psychiatric illness that hinders adherence to the protocol, such as psychosis, obsessive-compulsive neurosis, bipolar disorder treatment, diseases that require treatment with lithium, and suicide thoughts in the last 5 years prior to inclusion.
* Presence of neurological disease, liver disease or kidney disease (diseases which have led to hospitalization or prolonged treatment).
* History of sickle cell anemia.
* Asplenia (no spleen or its removal).
* History of alcohol use/abuse (CAGE criterion) or illicit drugs.
* Blood pressure above 140/90 mmHg at screening or hypertension requiring drug treatment.
* Coagulopathy diagnosed by a doctor or report of capillary fragility (eg, bruising, bleeding, etc.) after injections or blood sampling.
* Active malignancy (eg, any type of cancer) or treated so it may relapse during the study.
* History of allergy to vaccines containing adjuvants composed of lipids (GLA or MPL)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Safety of the vaccine | 4 months after the first dose
  Safety and tolerability of the vaccine (sm14 antigen plus GLA adjuvant) against schistosomiasis in health adults

SECONDARY OUTCOMES:
Proportion of seroconversion | 30 days after the third vaccine dose
  Proportion of seroconversion for sm14 antigen 30 days after the complete vaccinal schedule (3 doses, 30 days apart)
Cellular immune response to sm-14 vaccination in health adults | 30 days after the third vaccine dose
  Determine the cellular immune responses and their correlation to the development and magnitude of humoral responses

CONTACTS AND LOCATIONS:
Overall Officials: Marilia S Oliveira, MD, MsC, Principal Investigator — Instituto de Pesquisa Clínica Evandro Chagas (IPEC)
Locations (1):
- Instituto de Pesquisa Clínica Evandro Chagas (IPEC) - Fiocruz, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Santini-Oliveira M, Coler RN, Parra J, Veloso V, Jayashankar L, Pinto PM, Ciol MA, Bergquist R, Reed SG, Tendler M. Schistosomiasis vaccine candidate Sm14/GLA-SE: Phase 1 safety and immunogenicity clinical trial in healthy, male adults. Vaccine. 2016 Jan 20;34(4):586-594. doi: 10.1016/j.vaccine.2015.10.027. Epub 2015 Nov 10. PMID 26571311